CLINICAL TRIAL: NCT02540889
Title: Listen-In: the Development and Testing of a Web-based Therapy Application for Patients With Impaired Speech Comprehension Caused by Stroke
Brief Title: Listen in: Developing and Testing a Therapy Application for Patients With Speech Comprehension Deficits After Stroke.
Acronym: Listen-in
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14/0452
Record Dates: First submitted 2015-08-28; First posted 2015-09-04 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2017-07

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trial arm (Experimental): 100 hours of therapy.
  Interventions: Behavioral: Auditory comprehension therapy.
- Normal therapy arm (No Intervention): 12 weeks of normal therapy.

INTERVENTIONS:
Behavioral: Auditory comprehension therapy. — 100 hours of Auditory comprehension therapy embedded within a computer game.
  Arms: trial arm

SUMMARY:
The main aim is to develop and test the clinical efficacy of a novel, web based, rehabilitation application. Listen-In will provide an effective speech comprehension training tool that patients with aphasia can use to practice independently. This will free up therapists time to provide additional assessment, supervision and functional intervention in a highly cost effective manner.

DETAILED DESCRIPTION:
The main aim is to develop and test the clinical efficacy of a novel, web based, rehabilitation application. Listen In will provide an effective speech comprehension training tool that patients can use to practice independently. This will free up SALT time to provide additional assessment, supervision and functional intervention in a highly cost effective manner.

Phase 1 (24 months. London, Newcastle, Cambridge): Development of Listen In, including diagnostic and therapeutic components, driven by patient user's feedback (alpha and beta testing). The intervention is detailed below and is based on current SALT practice. It will be adaptive, provide feedback and target auditory perception at many levels: the phonemic, lexical and sentence level processing of heard verbal stimuli, as well as auditory short term memory and nonverbal sound discrimination.

Phase 2 (12 months. London and Cambridge): A pilot, randomised, crossover, clinical trial of Listen-In in a group of aphasic patients in the chronic post-stroke period. A power calculation suggests that we will need 36 patents, 18 in each arm. The comparison will be standard SALT clinical care. The main outcome measure is a clinically relevant improvement on the comprehension of spoken language score of the Comprehensive Aphasia Test (Swinburn, 2004). Secondary outcomes include improvements in social activity and participation. The milestones for this phase will be: 50% recruitment into study and last patient, last visit.

Phase 3 (funded outside i4i grant) will be the rollout of the therapy application on the internet with a pragmatic trial of whether therapy gains can be made outside the confines of a clinical trial. The comparison will be on similar outcome measures as Phase 2 with a control test on sustained attention (internal control) that we predict will not improve with therapy.

ELIGIBILITY:
Inclusion Criteria:

* any type of stroke but greater than 6 months post onset
* evidence of receptive aphasia
* English as their main language
* able to give informed consent
* age 18 years or above
* no diagnosis of degenerative brain disease.

Exclusion Criteria:

* Stroke less than 6 months post onset
* No evidence of receptive aphasia
* English not their main language
* Unable to give informed consent
* Less than 18 years old
* diagnosis of degenerative brain disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Improvement in auditory comprehension on the comprehensive aphasia test. | Measured over 36 weeks (0,12,24,36) weeks
  Investigation of improvement on a functionally relevant area of a widely used test of aphasia.

SECONDARY OUTCOMES:
Improvement in functional communication | Measured over 36 weeks (0,12,24,36) weeks
  Using patient reported outcomes to look at functional communication changes.
Improvement in production of language | Measured over 36 weeks (0,12,24,36) weeks
  Investigation of improvement on a functionally relevant area of a widely used test of aphasia.
Performance on the Sustained attention to response task | Measured over 36 weeks (0,12,24,36) weeks
  Investigation of improvement on sustained attention using the SART.
Environmental sounds test | Measured over 36 weeks (0,12,24,36) weeks
  Investigation of improvement on the non verbal environmental sounds test.
Test of semantics | Measured over 36 weeks (0,12,24,36) weeks
  Investigation of improvement in semantics knowledge.
Improvement in written language comprehension | Measured over 36 weeks (0,12,24,36) weeks
  Investigation of improvement on a functionally relevant area of a widely used test of aphasia.
Improvement on auditory descrimination | Measured over 36 weeks (0,12,24,36) weeks
  Investigation of improvement on a test of auditory discrimination developed by Dr Holly Robson.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Leff, PhD, Principal Investigator — ucl
Locations (1):
- UCLondon, London, United Kingdom

REFERENCES:
- [Derived] Fleming V, Brownsett S, Krason A, Maegli MA, Coley-Fisher H, Ong YH, Nardo D, Leach R, Howard D, Robson H, Warburton E, Ashburner J, Price CJ, Crinion JT, Leff AP. Efficacy of spoken word comprehension therapy in patients with chronic aphasia: a cross-over randomised controlled trial with structural imaging. J Neurol Neurosurg Psychiatry. 2020 Nov 5;92(4):418-24. doi: 10.1136/jnnp-2020-324256. Online ahead of print. PMID 33154182